CLINICAL TRIAL: NCT02676700
Title: The Effect of Pelvic Floor Muscle Training With or Without Kaatsu Training for Women With Stress Urinary Incontinence
Brief Title: Pelvic Floor Muscle Training and Kaatsu Training for Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Ulla Due, Physiotherapist, M.Sc, Ph.D., Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2013-125
Record Dates: First submitted 2016-01-31; First posted 2016-02-08 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Urinary Stress Incontinence
Keywords: Urinary stress incontinence; pelvic floor muscle; Kaatsu training
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pelvic floor muscle training and Kaatsu (Active Comparator): Participants are instructed in the PFMT program by primary investigator and instructed in Kaatsu training by a research nurse. The Kaatsu training is performed 4 times a week before PFMT. The program includes 2 x 15 knee extensions with partly occlusion of the blood supply to the thigh. Training level is >12 RM. Training is performed sitting on a chair and rubber bands are used to increase resistance. Training adherence and bother with the training is reported in a training diary. At week 6 the research nurse adjusts the training program.
  The PFMT program includes three sets of 10 contractions with an intensity of >12 RM and is to be performed 4 times a week.
  Training adherence and any bother with the training is reported in a training diary.
  Interventions: Behavioral: Pelvic floor muscle training and Kaatsu
- pelvic floor muscle training (Active Comparator): Participants perform the same PFMT program as the intervention group. The PFMT program includes three sets of 10 contractions with an intensity of >12 RM and is to be performed 4 times a week.
  Training adherence and any bother with the training is reported in a training diary.
  Interventions: Behavioral: Pelvic floor muscle training

INTERVENTIONS:
Behavioral: Pelvic floor muscle training and Kaatsu — The intervention includes three outpatient visits (weeks 0, 6 and 12) and between visits the participants perform PFMT and Kaatsu training as home training
  Arms: Pelvic floor muscle training and Kaatsu
Behavioral: Pelvic floor muscle training — The intervention includes three outpatient visits (weeks 0, 6 and 12) and between visits the participants perform PFMT as home training
  Arms: pelvic floor muscle training

SUMMARY:
This study examines the effect of adding so called Kaatsu training to pelvic floor muscle training. Half the participants will perform Kaatsu training on their thigh muscles followed by pelvic floor muscle training. The other half will receive pelvic floor muscle training alone.

DETAILED DESCRIPTION:
Stress urinary incontinence (SU) is a common problem among adult women . Pelvic floor muscle training (PFMT) is recommended as first line treatment but PFMT is not always efficient and some women cannot comply with the intensive PFMT needed to obtain effect because of weakened or damaged muscles caused by vaginal delivery and age related changes.

Hypothetically alternative methods could be used to enhance the effect of a strength-training program. A low intensity training program with a simultaneous partial occlusion of the blood supply for the training muscle, so called "Kaatsu" training has been found to increase muscle strength faster than ordinary strength training but with much less effort. It seems difficult to make occlusion of the pelvic floor muscles during PFMT but a study found that low intensity training of the quadriceps femoris with partial occlusion of the blood supply did not only increase muscle strength of the quadriceps femoris muscle but also of the biceps humeri muscle if that muscle was trained with low-load training and no occlusion in the same training session. The specific reason for this this "cross-transfer effect" could not be fully explained but it was believed to be caused by a systemic effect caused by growth hormones. The aim of this study is therefore to examine if Kaatsu training offered in relation to a low-load PFMT program can increase the effect of PFMT in women with SUI

ELIGIBILITY:
Inclusion Criteria:

* ICIQ-SF ≥ 12
* Urinary stress incontinence
* Ability to contract pelvic floor muscles
* Normal bladder capacity and normal flow during micturition with at least one micturition of > 350 ml

Exclusion Criteria:

* Urgency urinary incontinence
* Cognitive problems
* Physical inability to perform Kaatsu program
* Inability to understand and read Danish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02; Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
ICIQ-SF (International Consultation on Incontinence Questionnaire - Short Form ) | 12 weeks
  Subjective measure of severity of urinary loss and impact on quality of life

SECONDARY OUTCOMES:
ICIQ-SF | 6 weeks
  Subjective measure of severity of urinary loss and impact on quality of life
UPR (Urethral Pressure Reflectometry) | 12 weeks
  UPR is a novel method measuring the pressure and the cross-sectional area of the female urethra. The difference in urethral opening pressure during pelvic floor muscle contraction before and after intervention is measured in cm H2O
PGI-I (Patient Global Index of Improvement scale) | 6 and 12 weeks
  Global scale
Three days bladder diary | 6 and 12 weeks
  Diary to report number of incontinence episodes
VAS (Visual Analog Scale) | 6 and 12 weeks
  Scale used to report bother with performing the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Due, PT, Ph.D, Principal Investigator — Department of Gynecology and Obstetrics, Herlev-Gentofte Hospital; Soren Gräs, MD, Study Director — Department of Gynecology and Obstetrics, Herlev-Gentofte Hospital; Niels Klarskov, MD, lecturer, Study Director — Department of Gynecology and Obstetrics, Herlev-Gentofte Hospital; Anders Vinther, PT, Ph.D., Study Director — Herlev-Gentofte hospital; Gunnar Lose, MD, Prof, Study Director — Department of Gynecology and Obstetrics, Herlev-Gentofte Hospital
Locations (1):
- Department of Gynecology and Obstetrics, Herlev-Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madarame H, Neya M, Ochi E, Nakazato K, Sato Y, Ishii N. Cross-transfer effects of resistance training with blood flow restriction. Med Sci Sports Exerc. 2008 Feb;40(2):258-63. doi: 10.1249/mss.0b013e31815c6d7e. PMID 18202577